CLINICAL TRIAL: NCT00135031
Title: A Multicenter, Double-Blind, Randomized, Placebo-Controlled, Dose-Ranging Safety and Efficacy Evaluation of Bifidobacterium Infantis 35624 in Female Subjects With Irritable Bowel Syndrome
Brief Title: Efficacy of an Encapsulated Probiotic Bifidobacterium Infantis 35624 in Irritable Bowel Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Collaborators: Alimentary Health Ltd (Industry)
Responsible Party: Linda McKean, Procter & Gamble
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2002089
Record Dates: First submitted 2005-08-23; First posted 2005-08-25 (Estimated); Last update posted 2011-06-15 (Estimated); Status verified 2011-06

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Bifidobacterium infantis 35624

SUMMARY:
The purpose of this study was to determine the dose-ranging efficacy and safety profile of encapsulated Bifidobacterium infantis 35624 in female subjects with irritable bowel syndrome (IBS).

DETAILED DESCRIPTION:
The pathogenesis of irritable bowel syndrome (IBS) may have a a post-infectious inflammatory component, suggesting that altered gut bacterial flora are of relevance and that probiotics may be beneficial. This clinical trial examined the efficacy of an encapsulated probiotic in subjects with Rome II IBS. After a 2 week baseline, 362 female subjects were randomized to placebo or one of three doses of B. infantis 35624 once daily for 4 weeks. IBS symptoms were monitored daily and scored according to a 6-point Likert scale; stool frequency and form were also monitored daily. The primary efficacy variable was the abdominal pain score; secondary efficacy variables included other IBS symptom relief and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Meet Rome II criteria for the diagnosis of IBS
* Refrain from using probiotic supplements during the trial

Exclusion Criteria:

* Organic diseases, including inflammatory bowel disease, and significant systemic diseases
* Subjects over 55 years of age that had not had a sigmoidoscopy or colonoscopy performed in the previous five years
* Use of anti-psychotic medications within the prior three months
* Had major psychiatric disorder (DSM-II-R or DSM-IV), including major depression, psychoses, alcohol or substance abuse, within the past two years
* Were pregnant or nursing
* Had known lactose intolerance or immunodeficiency
* Had undergone any abdominal surgery, with the exception of hernia repair or appendectomy

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 362
Dates: Start 2004-01; Primary Completion 2004-09 (Actual); Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
The primary efficacy variable was the abdominal pain score

SECONDARY OUTCOMES:
Bloating/distension, sense of incomplete evacuation, straining, urgency, passage of gas, number of bowel movements, passage of mucus, a composite symptom score, subject's assessment of IBS symptom relief, and quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Peter J. Whorwell, M.D., Principal Investigator — Department of Medicine, Education and Research Centre, Wythenshawe Hospital, Manchester M23 9LT UK
Locations (20):
- United Kingdom (20):
  - The Orchard Medical Centre, Bristol, Bristol
  - Yaxley Group Practice, The Health Centre, Peterborough, Cambridgeshire
  - The Staploe Medical Centre, Soham, Cambridgeshire
  - Wansford Surgery, Wansford, Cambridgeshire
  - Old School Surgery, Greenisland, County Antrim
  - Springhill Surgery, Bangor, County Down
  - Downpatrick Health Centre, Downpatrick, County Down
  - Little Common Surgery, Bexhill-on-Sea, East Sussex
  - Sea Road Surgery, Bexhill-on-Sea, East Sussex
  - Valleyfield Health Centre, High Valleyfield, Fife
  - Stanwell Road Surgery, Ashford, Middlesex
  - Belmont Health Centre, Harrow, Middlesex
  - The Frome Medical Practice, Frome, Somerset
  - The Burns Practice, Doncaster, South Yorkshire
  - The Burngreave Surgery, Sheffield, South Yorkshire
  - The Medical Centre, East Horsley, Surrey
  - The Penylan Surgery, Cardiff, Wales
  - Sherbourne Medical Centre, Royal Leamington Spa, Warwickshire
  - Hathaway Surgery, Chippenham, Wiltshire
  - Swindon Medical Research Centre, Abbeymeads Medical, Swindon, Wiltshire